CLINICAL TRIAL: NCT03032458
Title: Efficacy of Pethidine, Ketorolac And Xylocaine Gel As Analgesics For Pain Control In Shockwave Lithotripsy Single Blinded Randomized Controlled Trial
Brief Title: Efficacy of Pethidine, Ketorolac And Xylocaine Gel As Analgesics For Pain Control In Shockwave Lithotripsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD/16.11.72
Record Dates: First submitted 2017-01-10; First posted 2017-01-26 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Analgesia; Urolithiasis
Keywords: Shock Wave Lithotripsy; Ketorolac; Xylocaine Gel; Pethidine
MeSH Terms: conditions — Agnosia; Urolithiasis | interventions — Meperidine; Ketorolac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pethidine (Active Comparator): Pethidine 25 mg IV bolus (Pethidine hydrochloride 50mg ampule, Roche Pharmaceutical Company - Egypt)
  Interventions: Drug: Pethidine
- Ketorolac (Active Comparator): Ketolac 30 mg (ketorolac, Amriya Pharmaceutical Industries - Egypt)
  Interventions: Drug: Ketorolac
- Xylocaine Gel (Active Comparator): Xylocaine gel (lidocaine 2%, AstraZeneca Pharmaceutical Company - Egypt)
  Interventions: Drug: Xylocaine Gel

INTERVENTIONS:
Drug: Pethidine — pethidine 25 mg IV bolus injection before start of session plus placebo gel then then IV infusion, so that the total dose doesn't exceed 1mg/kg
  Other Names: Pethidine 50
  Arms: Pethidine
Drug: Ketorolac — ketorolac IV bolus injection before start of session plus placebo gel then 30 mg IV infusion so that total dose doesn't exceed 60 mg.
  Other Names: Ketolac
  Arms: Ketorolac
Drug: Xylocaine Gel — Xylocaine gel locally 15 minutes before session with 10 mg normal saline IV bolus before session then IV normal saline infusion then
  Other Names: lidocaine 2%
  Arms: Xylocaine Gel

SUMMARY:
A randomised prospective trial comparing the efficacy of pethidine, Ketorolac, and Xylocaine gel as analgesics for pain control in shockwave lithotripsy.

DETAILED DESCRIPTION:
Pain perception during shockwave lithotripsy (SWL) is affected by patient-related factors like age, gender, and body habitus moreover, young female patients, anxious and depressed patients or thin patients experience more pain during SWL.

Several physical variables influencing treatment-related pain have been identified: the type of the shockwave source, size, and site of stone burden, peak pressure of the shockwaves, diameter of the focal zone, and size of the aperture of the shockwave source reflecting the area of shockwave entry at the skin.

Pain relief during SWL is vital, not only to maintain patient comfort and satisfaction, but also to facilitate stone imaging and targeting by reducing patients' movements during successive shock wave impacts. Reduced patient movement enables increase fragmentation efficiency and reduce the risk of procedure-related morbidity. So, a relaxed, cooperative patient during treatment is paramount in maintaining stone targeting for optimal fragmentation.

Across 21 centers in the United Kingdom (UK), 17 distinct analgesia regimens were reported in SWL analgesia practice.

In 2016 European Association of Urology (EUA) guidelines for SWL Pain control stated that pain control during SWL is necessary to limit pain induced movements and excessive respiratory excursions, However no recommendation for proper analgesia in contrast to clear recommendation for Pain relief in patients with an acute stone episode.

The investigators will try in this trial to identify the best efficacious type of analgesia for patient during SWL in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal and upper ureteral stones amenable to SWL.

Exclusion Criteria:

* Allergy to pethidine.
* Allergy to Ketorolac.
* Allergy to Xylocaine gel.
* American Society of Anesthesiologists score ≥ 3 (ASA III or more).
* Pregnancy.
* Patients with a pacemaker.
* Bleeding diatheses.
* Uncontrolled urinary tract infection (UTI).
* Severe obesity which prevent targeting of the stone.
* Body Mass IndexBMI (40 or more)
* Arterial aneurysm in the vicinity of the stone.
* Anatomical obstruction distal to the stone.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Pain control __ Outcome Measure by "pain assessment scales of The National Initiative on Pain Control™ (NIPC™)" | 10 months

SECONDARY OUTCOMES:
Effect of anxiety on success of SWL __ Outcome Measure by "Generalized Anxiety Disorder 7-item " | 10 months
Effect of anxiety on success of SWL __ Outcome Measure by "The Patient Health Questionnaire (PHQ-9)" | 10 months
Compare stone free rate __ Outcome Measure by "ultrasound and plain x-ray" 1 week after session. If no residual stone, NCCT scan. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abol-Enein, MD, Phd, Study Chair — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Hassan Abol-Enein, MD, Phd (Study Chair) or Prof. Khaled Z. Sheir, MD ( Study Central Contact Backup)